CLINICAL TRIAL: NCT00489905
Title: Evaluation of Zoledronic Acid to Prevent Bone Loss in Men Receiving Androgen Deprivation Therapy for Prostate Cancer
Brief Title: Study on Evaluation of Zoledronic Acid to Prevent Bone Loss in Men Receiving Androgen Deprivation Therapy for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Baxter Healthcare Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2005.137-T; HARECCTR0500010
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Prostatic Neoplasms; Bone Density
Keywords: prostate cancer; bone mineral density
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zolderonic acid (Zometa)

SUMMARY:
The purpose of this study is to assess the effect of zoledronic acid on bone mineral density in prostatic cancer patients currently receiving androgen deprivation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients aged between 50-80 who is having or will have ADT. Baseline BMD in between -2 standard deviation (SD) and mean of that among young adults.

Exclusion Criteria:

* Patients with renal or liver problems, on calcium or other bisphosphonate therapy within six months before enrolling into the study.

Patients who have:

* Serum creatinine levels >212 µmol/L (2.4 mg/dL).
* Creatinine clearance <50 ml/min.
* WBC <4.0x109/L, Hgb <10 g/dL, platelets <140x109/L. Patients with known hypersensitivity to bisphosphonates. Patients with history of diseases with influence on bone metabolism, such as Page's disease of bone, primary hyperparathyroidism or osteoporosis.

Ages: 50 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-04; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Bone mineral density of lumber spine | 12 months after administration of zolderonic acid
Bone mineral density of femoral neck | 12 months after administration of zolderonic acid

SECONDARY OUTCOMES:
Change in serum creatinine, calcium, phosphate and alkaline phosphatase | From time of enrollment to 3 months after the last intervention
Change in creatinine clearance | From time of enrollment to 3 months after the last intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, Dr, Principal Investigator — Department of Surgery, Division of Urology, The Chinese University of Hong Kong
Locations (1):
- Department of Urology, Prince of Wales Hospital, Hong Kong, China